CLINICAL TRIAL: NCT04627753
Title: Phase II Study of Lenalidomide/Rituximab Maintenance for Transplantation Ineligible Patients With Primary CNS Diffuse Large B-cell Lymphoma (Nickname: Lemon-C Study)
Brief Title: Study of Lenalidomide/Rituximab Maintenance for Transplantation Ineligible Patients With PCNSL.
Acronym: Lemon-C
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kim, Seok Jin (Other)
Collaborators: Celltrion (Industry); Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor-Investigator, Kim, Seok Jin, MD, PhD, Division of hematology-oncology, Department of medicine, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-10-081
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Primary CNS Lymphoma
MeSH Terms: interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenalidomide and Rituximab therapy (Experimental): The clinical trial drug is administered in one cycle for 28 days and is administered as follows.
  Drug : Rituximab It will be administered 375 mg/m² IV infusion Day 1. (Rituximab: up to 6 cycles)
  Drug : Lenalidomide It will be administred 20 mg PO day 1 -21.
  The medication is taken for up to 2 years, and if there is no recurrence, it is stopped after 2 years
  , Or stop when disease progression is confirmed during the administration period.
  Interventions: Drug: Rituximab, lenalidomide

INTERVENTIONS:
Drug: Rituximab, lenalidomide — Maintenance for 2 years
  Other Names: Truxima Inj; Lenalid

SUMMARY:
* After standard treatment of primary central nervous system lymphoma (PCNSL), high-dose methotrexate induction therapy, and consolidation therapy, most patients reach complete remission, but within the first 6 months, 35-60% of patients refractory to treatment or experience relapse during the first treatment.
* The progression-free survival (PFS) period of relapsed patients is 2.2 months (0-29.6 months), and the survival period is reported as 3.5 months (0-29.6 months). After relapse, the majority of patients die within 2-4 months due to neurologic deterioration
* Consolidation therapy after induction therapy includes whole-brain radiation therapy, high-dose chemotherapy followed by autologous hematopoietic stem cell transplantation (auto-SCT), and high-dose chemotherapy alone.
* However, the median age of the inducing patient is 65 years, and more than half of the patients who are unable to transplant autologous hematopoietic stem cells (auto-SCT) after induction therapy account for more than half.
* Therefore, we intend to conduct a study to evaluate the efficacy and safety of maintenance therapy for rituximab and lenalidomide as one of the consolidation therapies for patients with primary central nervous system lymphoma (PCNSL).

DETAILED DESCRIPTION:
-As described, standard treatment for patients with primary central nervous system lymphoma is not yet based on a high level of evidence, and studies on consolidation therapy for elderly patients who cannot transplant this disease are very limited. Based on the Korea National Cancer Incidence Database, about 100 to 150 cases of primary central nervous system lymphoma are diagnosed per year in Korea, and 15 to 30% of them are judged to experience recurrence.

Rituximab and lenalidomide (RR) are drugs that are expected to play a role in patients with primary central nervous system lymphoma who have already refractory or relapsed as described above, but there is a big hurdle that the number of patients is limited. Since then, it has not been studied as consolidation therapy in elderly or non-transplantable patients. Therefore, the present investigators attempted to confirm the efficacy and safety of lenalidomide/rituximab maintenance therapy in patients with primary central nervous system lymphoma who received high-dose methotrexate-containing anticancer drug, but could not receive consolidation therapy with autograft.

ELIGIBILITY:
Inclusion Criteria:

1. Those who have been diagnosed with histopathological primary central nervous system lymphoma and who have completed standard chemotherapy for induction of remission of primary central nervous system lymphoma have reached a complete or partial response.
2. Those who are unable to transplant autologous hematopoietic stem cells for the following reasons

   * If you are 65 years of age or older or if you are judged to have a weak systemic condition before receiving high-dose chemotherapy
   * Refusal of autologous hematopoietic stem cell transplantation after high-dose chemotherapy
3. Adequate laboratory functional values

   * Absolute neutrophil count ≥ 1000/ul
   * Platelet count ≥ 50,000/ul
   * Hemoglobin ≥ 9.0 g/dL
   * Serum calcium ≤ 12.0mg/dL
   * Serum creatinine ≤ 1.5 X UNL
   * AST/ALT ≤ 2.5 X UNL
   * Total bilirubin ≤ 1.5 X UNL
4. Hepatitis B patients with combination of prophylactic antiviral therapy
5. ECOG PS 0-2
6. Those who can take oral medication
7. Written informed consent under institutional guidelines.
8. Female patients of child-bearing potential (FCBP) must have two negative pregnancy tests (sensitivity of at least 25 mIU/mL) prior to starting lenalidomide. The first pregnancy test must be performed within 10 to 14 days prior to the start of lenalidomide, and the second pregnancy test must be performed within 24 hours prior to the start of lenalidomide.
9. Effective method of contraception should be used during and for 28 days following the last dose of the drug

   - FCBP is defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
10. Male patients must use an effective barrier method of contraception during study and 28 days following the last dose if sexually active with a FCBP.

Exclusion Criteria:

1. If autotransplantation is planned after chemotherapy
2. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within six months prior to 1st day of 1st cycle.
3. Acute active infection requiring systemic antibiotics, antiviral (except antiviral therapy directed at hepatitis B) or antifungal agents.
4. Uncontrolled hepatitis C infection and/or hepatitis B (except for patients with hepatitis B surface antigen [SAg] or core antibody receiving and responding to antiviral therapy directed at hepatitis B: these patients are allowed).
5. . Known human immunodeficiency (HIV) seropositive
6. Those who are unable to take oral medication
7. Patients with a history of malignant tumors other than the target diseases except for the following cases

   * If the tumor has not been treated for at least 5 years or is disease-free
   * Patients at least 1 year after complete resection of basal cell carcinoma / squamous cell carcinoma or successful treatment of cervical epithelial cancer
8. Adverse reactions within 30 days prior to screening Severe gastrointestinal bleeding exceeding Grade 2 according to the Common Terms Criteria 4.03 version criteria
9. Occurrence of blood clots or embolism within 6 months before starting screening
10. Patients with hypersensitivity to THIS DRUG and other ingredients of THIS DRUG (e.g., angioedema, Stevens-Jones syndrome, toxic epidermal necrosis, etc.)
11. Patients with seizure disorder requiring medication
12. Female patients who are pregnant or lactating.
13. Patients with genetic problems such as galactose intolerance, lapp lactase deficiency, or glucose-galactose malabsorption.
14. Patients with hyperreactivity to rituximab.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-11-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
1 year progression free survival | 12 months
  The incidence of tumor progression or death from all causes during the 1-year follow-up period from the first drug administration date.

SECONDARY OUTCOMES:
2-year progression free survival | 24 months
  The incidence of tumor progression or death from all causes during the 2-year follow-up period from the first drug administration date.
Overall survival | 24 months
  The time from the first drug administration to death from any cause.
Overall response | 24 months
  The proportion of patients who achieve complete and partial response.
Toxicity profiles | from the date of informed consent signature to 30 days after last drug administration.
  Clinical and laboratory toxicity/symptomatology will be graded based on the NCIC CTG v4.03. Adverse events not reported in NCIC CTG will be categorized into mild, moderate, severe, and fatal and further classified to CTCAE Grades 1-4.

CONTACTS AND LOCATIONS:
Overall Officials: Seok Jin Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea